CLINICAL TRIAL: NCT00005767
Title: Dynamic Aspects of Amino Acid Metabolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR00109-0740; M01RR000109 (NIH)
Record Dates: First submitted 2000-06-01; First posted 2000-06-02 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Kidney Diseases
Keywords: Amino Acid Metabolism
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Cross-Sectional

SUMMARY:
This protocol seeks to define aspects of intestinal and hepatic uptake and metabolism of several amino acids. The major hypothesis to be tested is that the splanchic bed (intestine and liver) conserves essential amino acids and metabolites while synthesizing and metabolizing nonessential amino acids. The aims of the study include defining the relative roles of enteral and hepatic extraction/metabolism in the disposition of glutamate, alanine, methionine and other amino acids. Emphasis will also be placed on studies of the transamination of alpha-ketoisocaproic acid (KIC) to leucine since this reaction is of potential importance in the design of nutritional regimens for patients with renal disease.

ELIGIBILITY:
Inclusion Criteria:

* normal weight-for-height weight 50-80 kg
* normal physical activity
* no significant medical history
* healthy by medical exam and lab blood testing

Exclusion Criteria:

* subjects who exercise vigorously
* subjects who smoke

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States